CLINICAL TRIAL: NCT05342363
Title: Mechanical Cardiopulmonary Resuscitation During Treatment of Acute Respiratory Failure Through Extracorporeal Membrane Oxygenation.
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Physician, Goethe University
Other Study IDs: CPR during VV-ECMO
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Resuscitation; Venovenous Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardiopulmonary resuscitation during treatment with extracorporeal membrane oxygenation: Patients treated with venovenous extracorporeal membrane oxygenation (vv-ECMO) for acute respiratory distress syndrome (ARDS) during the retrospective observation period who required mechanical cardiovascular resuscitation (CPR) during their treatment.
- Treatment with extracorporeal membrane oxygenation without resuscitation: Patients treated with venovenous extracorporeal membrane oxygenation (vv-ECMO) for acute respiratory distress syndrome (ARDS) without the need for cardiovascular resuscitation during the retrospective observation period.

SUMMARY:
In-hospital cardiovascular arrest is associated with poor outcome despite prompt treatment and optimal on-site resources. The population of patients treated by venovenous extracorporeal membrane oxygenation (vv-ECMO) due to pulmonary failure is a very challenging group of patients. To date, the frequency, causes and outcome of cardiovascular arrest in these patients have not been studied. We are aiming to conduct a retrospective observational study of all vv-ECMO patients treated at our ARDS centre.

ELIGIBILITY:
Inclusion Criteria:

Patients treated with veno-venous extracorporeal membrane oxygenation (vv-ECMO) due to respiratory failure during acute respiratory distress syndrome (ARDS).

Exclusion Criteria:

Patients treated with veno-arterial extracorporeal membrane oxygenation (va-ECMO)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with veno-venous extracorporeal membrane oxygenation (vv-ECMO) for respiratory failure in acute respiratory distress syndrome (ARDS). And in addition required mechanical cardiovascular resuscitation treatment during existing therapy with veno-venous extracorporeal membrane oxygenation (vv-ECMO).
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Survival of mechanical cardiovascular resuscitation | During the intensive care stay ( usually between 2 and 8 weeks)
  Survival of mechanical cardiovascular resuscitation

SECONDARY OUTCOMES:
Incidence of cardiovascular resuscitation i | During the observation period 2019-2022
  Incidence of cardiovascular resuscitation in patients treated with venovenous extracorporeal membrane oxygenation.
Complications of resuscitation treatments | During the intensive care stay ( usually between 2 and 8 weeks)
  Complications of cardiovascular resuscitation in patients treated with venovenous extracorporeal membrane oxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
Sharing patient data with third parties is subject to national and local law restrictions and regrettably not possible.